CLINICAL TRIAL: NCT06265870
Title: Comparison of Outcome Between Specific Anthelminthic Treatment According to Test Results and Empirical Anthelminthic Treatment in Eosinophilic Patient
Brief Title: Specific Versus Empirical Anthelminthic Treatment in Eosinophilia
Acronym: Eosinophilia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Thareerat Ananchaisarp, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parasite in Eosinophilia
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Eosinophilia
Keywords: eosinophilia; anthelminthic drugs; empirical treatment; stool examination
MeSH Terms: conditions — Eosinophilia | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific anthelminthic (Active Comparator): Participants were asked to provide stool samples for three consecutive days for testing through microscopy, culture, and PCR to detect parasites.
  * This study will combine wet smear and Kato's thick smear methods, with duplicate samples collected from each stool specimen to maximize parasite detection. To ensure reliability, two experienced microscopists will independently examine all four slides, and an independent report generated. In cases of discrepant results, a third microscopist will arbitrate, and the final diagnosis determined by majority vote.
  * Stool culture will look for Strongyloides stercoralis and hookworm larvae.
  * Stool PCR: Targeted gene of 7 helminths will be amplified and detected by multiplex real-time PCR. The reaction will be dividing into three assays.
  Following the analysis of the stool samples, participants will receive specific anthelminthic treatment tailored to the results of the stool tests.
  Interventions: Drug: Ivermectin or albendazole
- Empirical anthelminthic (Placebo Comparator): Participants will receive an empirical anthelminthic regimen consisting of albendazole 400 mg twice a day for seven consecutive days. Following this treatment, a follow-up complete blood count (CBC) will be requested to assess responsiveness.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Participants receive empiric anthelminthic treatment which is albendazole 400 mg twice a day for seven consecutive days
  Arms: Empirical anthelminthic
Drug: Ivermectin or albendazole — Participants will receive specific anthelminthic treatment tailored to the results of the stool tests
  Arms: Specific anthelminthic

SUMMARY:
There are a few guidelines recommend about management of eosinophilia worldwide, most of guielines recommend a thorough history-taking and physical examination. Subsequently, investigations are requested based on suspected causes. In cases where parasite infection is suspected, particularly in developing countries, stool microscopy and serology are recommended. However, limitations such as low sensitivity of stool microscopy, the inconvenience of collecting multiple stool samples, and the high cost and unavailability of serology may arise. Consequently, some physicians opt for empiric anthelminthic regimens in managing eosinophilic patients, even without stool tests or if stool test results are normal. If subsequent complete blood count (CBC) results show a recovery of absolute eosinophil count, it is assumed that eosinophilia was caused by a parasite infection. While some studies demonstrate the efficacy and simplicity of this approach, there is a risk of overestimating parasite infection in eosinophilic patients, potential adverse drug reactions from unnecessary anthelminthic treatment, and the possibility of drug resistance due to inappropriate dosing. To address this gap, no study has yet compared the efficacy between specific anthelminthic treatment based on test results and empirical anthelminthic treatment in eosinophilic patients. Therefore, the investigators are conducting this study.

DETAILED DESCRIPTION:
Eosinophilia is defined as an absolute eosinophil count exceeding 500 cells per microliter, calculated by multiplying the white blood cell count by the percentage of eosinophils.

Cause of eosinophilia vary from mild to life-threatening disease. Prevalence of each cause of eosinophilia vary on study population, the most common etiology in developing country is parasite infection.

Stool microscopy can be conducted using various methods. The Kato-Katz technique, recommended by the WHO, exhibits a sensitivity of only 52.4 percent (95%CI = 47.6 - 57.1 percent). More sensitive methods for parasite detection in stool, such as stool culture or PCR, are not readily available and can be costly. In the intervention group of this study, the investigators employed three different parasite detection methods (stool microscopy, stool culture, and PCR) to enhance sensitivity in detecting parasites.

ELIGIBILITY:
Inclusion Criteria:

* Participants who come for check-ups at general practitioner, primary care unit, and Srivejchavat Premium Center have an absolute eosinophil count greater than 500 cells/microliter with a white blood cell count less than 10,000 cells/microliter.
* Age at least 18 years old
* Consent to participate in research

Exclusion Criteria:

* Having any characteristics that need urgent care 1.1 Having history of unintended significant weight loss is defined as the loss of body weight exceeding 10% within a span of six months without deliberate attention.

1.2 Physical examination revealed a body temperature equal to or greater than 37.8 degrees Celsius, lymphadenopathy or hepatosplenomegaly.

1.3 CBC revealed blast cell

* Receiving anthelminthic drug within 6 months
* Underlying cancer (active stage), HIV, HBV, HCV, collagen vascular disease, active TB
* Allergy to albendazole, ivermectin, or metronidazole
* Pregnancy or lactation
* Serum transaminase higher than 2 times of upper normal limit
* Taking medications that may induce eosinophilia within the past three months, such as herbal supplements, NSAIDs, Salicylic acid, Carbamazepine, Colchicine, Nitrofurantoin, Dapsone, or Minocycline, was reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Eosinophilia recovery | From receive anthelminthic treatment to the end of treatment at 4 weeks
  Recovery from eosinophilia was defined as an absolute eosinophil count of less than 500 cells per microliter, as measured from the complete blood count (CBC) four weeks after receiving anthelminthic treatment.

SECONDARY OUTCOMES:
Change in AEC | From receive anthelminthic treatment to the end of treatment at 4 weeks
  Comparing the change in AEC from baseline between the "specific treatment group" and the "empirical treatment group" using either a paired t-test or the Wilcoxon signed-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Thareerat Ananchaisarp, Principal Investigator — Prince of Songkla University - Hat Yai Campus: Prince of Songkla University
Locations (1):
- Prince of Songkla University - Hat Yai Campus: Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available at primary researcher and may share with author research on reasonable request.

REFERENCES:
- [Result] Chanswangphuwana C, Uaprasert N, Moonla C, Rojnuckarin P. Causes and outcomes of hypereosinophilia in a tropical country. Asian Pac J Allergy Immunol. 2024 Dec;42(4):403-408. doi: 10.12932/AP-221220-1021. PMID 33865302
- [Result] Ananchaisarp T, Chamroonkiadtikun P, Julamanee J, Perdvong K, Chimpalee T, Rattanavirakul N, Leelarujijaroen N, Hathaipitak T, Tantinam T. Prevalence and management of eosinophilia based on periodic health examinations in primary care clinics. Asian Biomed (Res Rev News). 2023 Jun 16;16(5):273-282. doi: 10.2478/abm-2022-0030. eCollection 2022 Oct. PMID 37551315
- [Result] Shomali W, Gotlib J. World Health Organization-defined eosinophilic disorders: 2022 update on diagnosis, risk stratification, and management. Am J Hematol. 2022 Jan 1;97(1):129-148. doi: 10.1002/ajh.26352. Epub 2021 Oct 8. PMID 34533850
- [Result] Butt NM, Lambert J, Ali S, Beer PA, Cross NC, Duncombe A, Ewing J, Harrison CN, Knapper S, McLornan D, Mead AJ, Radia D, Bain BJ; British Committee for Standards in Haematology. Guideline for the investigation and management of eosinophilia. Br J Haematol. 2017 Feb;176(4):553-572. doi: 10.1111/bjh.14488. Epub 2017 Jan 23. No abstract available. PMID 28112388
- [Result] Magnaval JF, Laurent G, Gaudre N, Fillaux J, Berry A. A diagnostic protocol designed for determining allergic causes in patients with blood eosinophilia. Mil Med Res. 2017 May 23;4:15. doi: 10.1186/s40779-017-0124-7. eCollection 2017. PMID 28546866
- [Result] Vaisben E, Brand R, Kadakh A, Nassar F. The role of empirical albendazole treatment in idiopathic hypereosinophilia - a case series. Can J Infect Dis Med Microbiol. 2015 Nov-Dec;26(6):323-4. doi: 10.1155/2015/531675. PMID 26744590
- [Result] Insiripong S, Siriyakorn N. Treatment of eosinophilia with albendazole. Southeast Asian J Trop Med Public Health. 2008 May;39(3):517-20. PMID 18564693
- [Result] Chen B, Fu Y, Wang Z, Rong Q, Zhang Q, Xie J, Kong X, Jiang M. Eosinophilia attention, diagnosis, treatment, and awareness in physicians: a cross-sectional survey. Ther Adv Chronic Dis. 2023 Jan 24;14:20406223221146938. doi: 10.1177/20406223221146938. eCollection 2023. PMID 36712467
- [Result] Kim DW, Shin MG, Yun HK, Kim SH, Shin JH, Suh SP, Ryang DW. [Incidence and causes of hypereosinophilia (corrected) in the patients of a university hospital]. Korean J Lab Med. 2009 Jun;29(3):185-93. doi: 10.3343/kjlm.2009.29.3.185. Korean. PMID 19571614
- [Result] Wardlaw AJ, Wharin S, Aung H, Shaffu S, Siddiqui S. The causes of a peripheral blood eosinophilia in a secondary care setting. Clin Exp Allergy. 2021 Jul;51(7):902-914. doi: 10.1111/cea.13889. Epub 2021 Jun 3. PMID 34080735
- [Result] Tefferi A, Patnaik MM, Pardanani A. Eosinophilia: secondary, clonal and idiopathic. Br J Haematol. 2006 Jun;133(5):468-92. doi: 10.1111/j.1365-2141.2006.06038.x. PMID 16681635
- [Result] Guo C, Bochner BS. Workup for eosinophilia. Allergy Asthma Proc. 2019 Nov 1;40(6):429-432. doi: 10.2500/aap.2019.40.4264. PMID 31690387
- [Result] Kuang FL. Approach to Patients with Eosinophilia. Med Clin North Am. 2020 Jan;104(1):1-14. doi: 10.1016/j.mcna.2019.08.005. PMID 31757229
- [Result] Rosenwasser LJ. Approach to patients with eosinophilia. Mo Med. 2011 Sep-Oct;108(5):358-60. PMID 22073495
- [Result] Simon D, Simon HU. Eosinophilic disorders. J Allergy Clin Immunol. 2007 Jun;119(6):1291-300; quiz 1301-2. doi: 10.1016/j.jaci.2007.02.010. Epub 2007 Apr 2. PMID 17399779
- [Result] Carranza-Rodriguez C, Escamilla-Gonzalez M, Fuentes-Corripio I, Perteguer-Prieto MJ, Garate-Ormaechea T, Perez-Arellano JL. Helminthosis and eosinophilia in Spain (1990-2015). Enferm Infecc Microbiol Clin (Engl Ed). 2018 Feb;36(2):120-136. doi: 10.1016/j.eimc.2015.11.019. Epub 2016 Jan 27. English, Spanish. PMID 26827134
- [Result] Khoury P, Bochner BS. Consultation for Elevated Blood Eosinophils: Clinical Presentations, High Value Diagnostic Tests, and Treatment Options. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1446-1453. doi: 10.1016/j.jaip.2018.04.030. PMID 30197068
- [Result] Khanna V, Tilak K, Mukhopadhyay C, Khanna R. Significance of Diagnosing Parasitic Infestation in Evaluation of Unexplained Eosinophilia. J Clin Diagn Res. 2015 Jul;9(7):DC22-4. doi: 10.7860/JCDR/2015/12222.6259. Epub 2015 Jul 1. PMID 26393130